CLINICAL TRIAL: NCT05828433
Title: Effectiveness of Epley-Canalith Repositioning Procedure Versus Vestibular Rehabilitation Therapy in Diabetic Patients With Benign Paroxysmal Positional Vertigo: A Randomized Trial
Brief Title: Effect of Epley-Canalith Repositioning Procedure and Vestibular Rehabilitation Therapy in Diabetic Patients With BPPV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Mohammad Abu Shaphe (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Mohammad Abu Shaphe, Associate Professor, University of Jazan
Organization: University of Jazan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04/JUREC/15PT.2022
Record Dates: First submitted 2023-03-21; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epley-Canalith Repositioning (Experimental): Step 1: The patient was brought down with the head tilted 45 degrees towards the af-fected canal as in Hallpike test. The neck was extended.
  Step 2: The head was rotated 90 degrees towards the unaffected side. The neck was extended.
  Step 3: The head and body were rotated by further 90 degrees from the previous positions (now face down). The neck was in neutral position.
  Step 4: The patient was brought into a sitting position while having their head turned constantly in the direction of the unaffected side.
  Step 5: The head was turn forward and the chin was kept 20° down for a minute
  Interventions: Other: Epley-Canalith Repositioning
- Vestibular Rehabilitation Therapy (Experimental): Habituation exercises Gaze stability exercises and balance training
  Interventions: Other: Vestibular Rehabilitation Therapy

INTERVENTIONS:
Other: Epley-Canalith Repositioning — Epley-Canalith Repositioning The intervention was given for approximately 15min, for 2 times in a week, for 4 weeks.
  Arms: Epley-Canalith Repositioning
Other: Vestibular Rehabilitation Therapy — Vestibular Rehabilitation Therapy Habituation exercises: The patients were asked to repeat the exercises 5 -10 times for 5 to 10 min, for 2 days in a week, for 4 weeks.
  Gaze stability exercises and balance training: The exercises were performed in 3 sets or 5 repetitions, for 2 days in a week, for 4 weeks.
  Arms: Vestibular Rehabilitation Therapy

SUMMARY:
Benign paroxysmal positional vertigo (BPPV) is a common inner ear disorder characterized by brief episodes of vertigo caused by changes in head position. The condition can cause significant func-tional impairment and reduced quality of life. BPPV is especially common among diabetic patients. The Epley-Canalith Repositioning Procedure (CRP) and Vestibular Rehabilitation Therapy (VRT) are two commonly used interventions for the treatment of BPPV. The objective of this paper is to determine the effective therapy among Epley-Canalith Repositioning Procedure and Vestibular Rehabilitation for improving balance and posture control in Diabetic patients with Benign Parox-ysmal Positional Vertigo. Thirty subjects with Diabetes Mellitus (Type 2) suffering from Benign Paroxysmal Positional Vertigo (BPPV) were recruited for the study and randomly assigned to groups A and B, underwent Canalith Repositioning Procedure and Vestibular Rehabilitation Therapy respectively. The outcome measures of the study were Vertigo Symptom Scale- Short Form (VSS-sf) score and Berg Balance Scale Form (BBS) score assessed at pre -treatment (pre) and 4 weeks post treatment (post).

DETAILED DESCRIPTION:
Research Objectives:To determine the effective therapy among Epley-Canalith Repositioning Procedure and Vestibular Rehabilitation for improving balance and posture control in Diabetic patients with Benign Paroxysmal Positional Vertigo

Methods: Thirty subjects were recruited for the proposed study on the basis of inclusion and exclusion criteria. Patients who are diagnosed with posterior canal BPPV by ENT physician and diabetes by the physician through laboratory investigations, both male and female aged between 20 to 70 years, Positive Dix -Hallpike test, Nystagmus lasting less than 60 seconds, willing to participate in the study and with a minimum score of 25/56 in Berg Balance Scale were included. Whereas, patients taking antivertigo drugs, who had been treated for similar vertigo experience, disease of different origin that may cause vertigo like migraine, multiple sclerosis, stroke, traumatic brain injury, if CRP has been done before, other causes of peripheral vertigo such as Meniere's disease, vestibular neuritis, labrynthitis and perilymphatic fistula, pathologies contraindicated for Dix- hallpike maneuver like prolapse intervertebral disk, cervical spine instability, cervical myelopathy, previous cervical spine surgery were excluded. Those meeting the criteria will be randomized into Group A i.e., Epley-Canalith Repositioning and Group B i.e., Vestibular Rehabilitation Therapy through lottery method.

Interventions In Group A (control group), the affected posterior canal (it is the posterior semi-circular canal of the under most ear when the classic nystagmus is provoked) was predetermined by Dix-Hallpike test. The time of latency and duration of induced nystagmus was recorded by an assistant using stopwatch. This provided an estimate of the time required for the canalith bolus trough 90°.

Procedure will be explained to the patients before the intervention. The patients will be asked to keep the eyes open to watch the nystagmus. The patient will be seated length wise on the examination table in search a way that when brought to the Hallpike position, the head should extend beyond the end of the table. An assistant was asked to stand by the side of affected canal.

Step 1: The patient was brought down with the head turned 45° towards the affected canal as in Hallpike test. The neck was extended.

Step 2: The head was rotated 90° towards the unaffected side. The neck will be extended Step 3: The head and body was rotated by further 9°0 from the previous positions (now face down). The neck was in neutral position. Step 4: The patient was brought up in siting position while the head was kept turning towards the unaffected side. Step 5: The head was turned forward and the chin will be kept 20° down for a minute.

Since all the patients were having nystagmus lasting for less than 60 seconds, each position was maintained for 60 second. The procedure will be repeated until no nystagmus will be observed during the last cycle or until no progress is apparent in the last two cycles.

The intervention will be given for approximately 15min, for 2 times in a week, for 4 weeks.

Before going home, all the patients were given instructions:

* The patients were asked to wait for 10 minutes after the maneuver is performed before going home
* Patients were instructed not to lie supine, to keep their head at 45 reclining positions while sleeping for 2 days.
* All patients were asked to avoid provoking head positions like bending over, looking up or down for 7 days following the procedure.

Group B received Vestibular Rehabilitation Therapy which consisted of habituation exercises, gaze stability and balance training. Habituation exercises: The patient were instructed to sit on the side the examining couch. Then he was warned that the exercises could worsen the frequency and intensity of vertigo in the beginning but that they should not alarmed because the symptoms would subside with the continuation of the intervention. In this testing, each maneuver is done in a passive way. For each measurement, it was noted whether vertigo is elicited (M+ or M-). Intensity and duration of vertigo will be recorded. When nystagmus is observed, its presence or absence is noted (Ny+ or Ny-). In case of exacerbation of symptoms, the exercises will be modified by decreasing the repetition or stopping the exercises until the symptoms disappeared. The frequency and duration of the exercises will be customized according the patient's response to the exercises. In this study, the patients were asked to repeat the exercises 5 -10 times for 5 to 10 min, for 2 days in a week, for 4 weeks. The exercises program were be graded so that the patient progresses from easily tolerated movements to difficult ones. Gaze stability exercises and balance training: The exercises were progressed from sitting to standing and support surface conditions were systematically varied progressing from firm surface to compliant and regular surfaces. The exercises were performed in 3 sets or 5 repetitions, for 2 days in a week, for 4 weeks. Data collection In this study, 30 subjects who fulfilled the inclusion criteria were included. Those meeting the criteria met with the physiotherapist who explained the project. Subjects were provided with the general guidance and information about the project and given time to consider involvement. The subjects will be given further opportunity to ask questions and then they will give a consent form.

After giving consent, patients were assessed with Dix- hallpike, Vertigo Symptom Scale -sf, Berg Balance Scale before the intervention and the findings will be recorded. The patients will be divided into 2 groups, Group A (N =15) and Group B (N=15). All the outcome were again recoded after the 4 weeks of intervention.

Data analysis Data was summarized as Mean ± SE (standard error of the mean). Pre and post groups were compared by paired t test. Pre to post change (pre-post or post-pre) in outcome measures of two independent groups will be compared by independent Student's t test. Discrete (categorical) data were summarized in number (n) and percentage (%) and compared by chi-square (χ2) test. A two-tailed (α=2) p<0.05 will be considered statistically significant. Analyses was performed on SPSS software (Windows version 17.0).

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with posterior canal BPPV by ENT physician
* Patients diagnosed with diabetes mellitus (Type 2) by the physician through laboratory investigations
* Both male and female
* Age between 20 to 70 years
* Positive Dix -Hallpike test
* Nystagmus lasting less than 60 seconds
* Willing to participate in the study
* Minimum score of 25/56 in Berg Balance Scale

Exclusion Criteria:

* Patients taking antivertigo drugs
* Treated for similar vertigo experience
* Disease of different origin that may cause vertigo like migraine, multiple sclerosis, stroke, traumatic brain injury
* CRP has been done before
* Other causes of peripheral vertigo such as Meniere's disease, vestibular neuritis, labyrinthitis and peri lymphatic fistula
* Pathologies contraindicated for Dix- Hallpike manoeuvre like prolapse inter-vertebral disk, cervical spine instability, cervical myelopathy
* Previous cervical spine surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-07 (Actual); Primary Completion 2023-01-17 (Actual); Study Completion 2023-01-17 (Actual)

PRIMARY OUTCOMES:
Vertigo symptom scale - short form | 4 weeks
  VSS consisting of 36 items addresses frequency and severity of dizziness symptoms within the last 12 months. Both a long (VSS-lf) and short a form (VSS-sf) is available. There are 15 items in the VSS-sf. The VSS-sf exhibits high internal consistency (alpha=0.9) and r=0.52 is the construct validity. It has high test -retest reliability is ICC VSS-sf = 0.88, VSS-V=0.90, VSS-A=0.90
Berg Balance Scale | 4 weeks
  It is used to test if a patient can securely balance himself while doing a series of prede-termined tasks. It consists of 14 items, each of which has a 5-point ordinal scale rang-ing from 0 to 4, with 0 denoting the lowest degree of function and 4 denoting the high-est level. The relative intra-rater reliability of the BBS with a pooled estimate of 0.98 (95% CI 0.97 to 0.99). Relative inter-rater reliability of the BBS with a pooled estimate of 0.97 (95% CI 0.96 to 0.98)

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No